CLINICAL TRIAL: NCT05503719
Title: Skin Closure With a Fast Absorbable Braided Suture Versus a Non-absorbable Monofilament Suture in Open Carpal Tunnel Release, a Randomized Controlled Trial
Brief Title: An Absorbable Suture Versus a Non-absorbable Suture in Carpal Tunnel Release, a Randomized Controlled Trial
Acronym: SUPER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KUH5203138
Record Dates: First submitted 2022-05-25; First posted 2022-08-17 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Carpal Tunnel Syndrome; Median Nerve Entrapment
Keywords: carpal tunnel; carpal tunnel syndrome; median nerve release; median nerve entrapment; surgery; suture; absorbable; non-absorbable
MeSH Terms: conditions — Carpal Tunnel Syndrome; Median Neuropathy

STUDY DESIGN:
Intervention Model Description: The participants are divided into two groups. The first group will get an absorbable suture and the second a non-absorbable suture.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Absorbable Suture (Experimental): Surgical wounds of this arm will be closed with an absorbable suture.
  Interventions: Procedure: Surgical wound closed with an absorbable suture
- Non-absorbable suture (Active Comparator): Surgical wounds of this arm will be closed with a non-absorbable suture.
  Interventions: Procedure: Surgical wound closed with a non-absorbable suture

INTERVENTIONS:
Procedure: Surgical wound closed with an absorbable suture — Patients undergoing median nerve release surgery will get their surgical wound closed with an absorbable suture according to their respective study group.
  Arms: Absorbable Suture
Procedure: Surgical wound closed with a non-absorbable suture — Patients undergoing median nerve release surgery will get their surgical wound closed with a non-absorbable suture according to their respective study group.
  Arms: Non-absorbable suture

SUMMARY:
The study compares two widely used treatments in closing the wound after open carpal tunnel release surgery: absorbable and non-absorbable sutures. It is conducted as a randomized controlled trial, where the participants are divided into two research groups. The visual outcome of the scar will be evaluated a year after the surgery.

DETAILED DESCRIPTION:
Absorbable sutures are more cost efficient and eliminate the need for suture removal both reducing costs and abolishing suture removal pain. We will study the difference in the visual outcome between the two groups. Based on former study the primary hypothesis is that there is no difference between the groups. The patients will evaluate their scars on a VAS-scale one year after the surgery. Secondarily we will focus on pain caused by the two sutures and take the suture removal pain into consideration. We expect therefore the non-absorbable suture to cause more pain in total. The evaluation will happen 2 weeks after the surgery by the patients.

ELIGIBILITY:
Inclusion Criteria

* carpal tunnel syndrome diagnosed with electro near my-graphs
* symptoms typical of carpal tunnel syndrome
* referral to carpal tunnel release
* informed consent signed
* the ability to receive the virtual questionnaire via email and answer it
* the ability to understand and answer the Finnish questionnaires

Exclusion Criteria

* repeat surgery
* known allergy to suture materials
* ongoing systemic steroid treatment
* ongoing chemotherapy
* ongoing immunomodulatory treatment
* past hypertrophic or keloid scars or other severe disturbances in wound healing
* age under 18, pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Visual outcome (VAS) of the scar (nice and ugly) as evaluated by the patient | 1 year
  The subjective aesthetics of the scar evaluated by the patient on a 10 cm visual analog scale (VAS) ranging from "the ugliest scar possible" to "the most beautiful scar possible". The proportion of ugly and nice scars will be reported. Outcome will be collected at one year time point.

SECONDARY OUTCOMES:
Visual outcome (VAS) of the scar (nice and ugly) as evaluated by an outcomes assessor | 1 year
  The subjective aesthetics of the scar evaluated by an outcome assessor on a 10 cm visual analog scale (VAS) ranging from "the ugliest scar possible" to "the most beautiful scar possible". The proportion of ugly and nice scars will be reported. Outcome will be collected at one year time point.
Pain (VAS) experienced by the patient from the sutures | 2 weeks
  The rate of any the pain in the area of the scar including pain related to possible suture removal evaluated by the patient on a 10 cm visual analog scale (VAS) ranging from "no pain at all" to "worst pain imaginable". Propotions of patients in ten groups from 0 to 10 will be reported. Outcome will be collected at two weeks time point.
The Boston Carpal Tunnel Questionnaire | 1 year
  A disease-specific measure of self-reported symptom severity and functional status measuring the effectiveness of the treatment. Outcome will be collected preoperatively and at one year time point.
The Net Promoter Score | 1 year
  Client experience, the likelihood of the patient to recommend the operation to a friend or a colleague
Costs | 1 year
  The mean difference between the two study arms in treatment costs.The required data will be analysed from the trial data and Finnish healthcare registries.
Adverse events | 1 year
  Adverse events will be monitored throughout the trial, and patients will be instructed to promptly report any potential serious adverse events. At the one-year follow-up point, the questionnaires will include an inquiry about whether the patient has experienced any adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital, Department of Orthopaedics, Traumatology and Hand Surgery, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: Yes
Pseudonymised patient-level data along with the study protocol, the informed consent form and the analytic code will be made available in case of a methologically sound proposal.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Anonymous patient level data will be available if the European Union regulations permit after the study has been finished. The end date is estimated to be 1 January 2027.
Access Criteria: Researchers who provide a methodologically sound proposal and reviewers of the journal where article will be published will be granted access. Proposals should be directed to aukusa@student.uef.fi. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Quinn JV, Wells GA. An assessment of clinical wound evaluation scales. Acad Emerg Med. 1998 Jun;5(6):583-6. doi: 10.1111/j.1553-2712.1998.tb02465.x. PMID 9660284
- [Background] Kundra RK, Newman S, Saithna A, Lewis AC, Srinivasan S, Srinivasan K. Absorbable or non-absorbable sutures? A prospective, randomised evaluation of aesthetic outcomes in patients undergoing elective day-case hand and wrist surgery. Ann R Coll Surg Engl. 2010 Nov;92(8):665-7. doi: 10.1308/003588410X12699663905113. Epub 2010 Jul 19. PMID 20659358
- [Background] Dosani A, Khan SK, Gray S, Joseph S, Whittaker IA. Clinical outcome and cost comparison of carpal tunnel wound closure with monocryl and ethilon: a prospective study. Hand Surg. 2013;18(2):189-92. doi: 10.1142/S0218810413500226. PMID 24164122
- [Background] Padua L, Coraci D, Erra C, Pazzaglia C, Paolasso I, Loreti C, Caliandro P, Hobson-Webb LD. Carpal tunnel syndrome: clinical features, diagnosis, and management. Lancet Neurol. 2016 Nov;15(12):1273-1284. doi: 10.1016/S1474-4422(16)30231-9. Epub 2016 Oct 11. PMID 27751557
- [Background] Van Spall HG, Toren A, Kiss A, Fowler RA. Eligibility criteria of randomized controlled trials published in high-impact general medical journals: a systematic sampling review. JAMA. 2007 Mar 21;297(11):1233-40. doi: 10.1001/jama.297.11.1233. PMID 17374817
- [Background] Zhang D, Earp BE, Blazar P. Evaluation and Management of Unsuccessful Carpal Tunnel Release. J Hand Surg Am. 2019 Sep;44(9):779-786. doi: 10.1016/j.jhsa.2019.05.018. Epub 2019 Jul 9. PMID 31300226
- [Background] Zhang D, Blazar P, Earp BE. Rates of Complications and Secondary Surgeries of Mini-Open Carpal Tunnel Release. Hand (N Y). 2019 Jul;14(4):471-476. doi: 10.1177/1558944718765226. Epub 2018 Mar 20. PMID 29557679
- [Background] Povlsen B, Tegnell I. Incidence and natural history of touch allodynia after open carpal tunnel release. Scand J Plast Reconstr Surg Hand Surg. 1996 Sep;30(3):221-5. doi: 10.3109/02844319609062819. PMID 8885019
- [Background] Atroshi I, Gummesson C, Johnsson R, Ornstein E, Ranstam J, Rosen I. Prevalence of carpal tunnel syndrome in a general population. JAMA. 1999 Jul 14;282(2):153-8. doi: 10.1001/jama.282.2.153. PMID 10411196
- [Background] Menovsky T, Bartels RH, van Lindert EL, Grotenhuis JA. Skin closure in carpal tunnel surgery: a prospective comparative study between nylon, polyglactin 910 and stainless steel sutures. Hand Surg. 2004 Jul;9(1):35-8. doi: 10.1142/s0218810404002017. PMID 15368623
- [Background] Erel E, Pleasance PI, Ahmed O, Hart NB. Absorbable versus non-absorbable suture in carpal tunnel decompression. J Hand Surg Br. 2001 Apr;26(2):157-8. doi: 10.1054/jhsb.2000.0545. PMID 11281671
- [Background] Kharwadkar N, Naique S, Molitor PJ. Prospective randomized trial comparing absorbable and non-absorbable sutures in open carpal tunnel release. J Hand Surg Br. 2005 Feb;30(1):92-5. doi: 10.1016/j.jhsb.2004.10.009. PMID 15620502
- [Background] Theopold C, Potter S, Dempsey M, O'Shaughnessy M. A randomised controlled trial of absorbable versus non-absorbable sutures for skin closure after open carpal tunnel release. J Hand Surg Eur Vol. 2012 May;37(4):350-3. doi: 10.1177/1753193411422334. Epub 2011 Oct 10. PMID 21987279
- [Background] Wang L. Guiding Treatment for Carpal Tunnel Syndrome. Phys Med Rehabil Clin N Am. 2018 Nov;29(4):751-760. doi: 10.1016/j.pmr.2018.06.009. Epub 2018 Sep 17. PMID 30293628
- [Background] Kim PT, Lee HJ, Kim TG, Jeon IH. Current approaches for carpal tunnel syndrome. Clin Orthop Surg. 2014 Sep;6(3):253-7. doi: 10.4055/cios.2014.6.3.253. Epub 2014 Aug 5. PMID 25177448
- [Background] Boya H, Ozcan O, Ozteki N HH. Long-term complications of open carpal tunnel release. Muscle Nerve. 2008 Nov;38(5):1443-1446. doi: 10.1002/mus.21068. PMID 18949783
- [Derived] Savolainen A, Nietosvaara Y, Sirola J, Hytonen M, Reito A, Heikkinen N, Raisanen MP. Skin closUre in carPal tunnEl Release (SUPER): protocol for a blinded randomised controlled trial comparing absorbable and non-absorbable sutures in carpal tunnel release. BMJ Open. 2024 Apr 16;14(4):e082289. doi: 10.1136/bmjopen-2023-082289. PMID 38626975